CLINICAL TRIAL: NCT04600635
Title: Effect of Confinement on Circadian Rhythms of Patients Integrated Into a Care Pathway for Bariatric Surgery
Acronym: CHRONO-CONF
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC20.281; 2020-A02212-37 (Other: ID RCB)
Record Dates: First submitted 2020-10-02; First posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with a medical history of obesity: Patients included are subject who entered a structured program of care for their obesity, with or without bariatric surgery.
  Interventions: Procedure: Bariatric surgery

INTERVENTIONS:
Procedure: Bariatric surgery — Some patients in the cohort are followed by a multidisciplinary team in preparation for bariatric surgery. Others have already undergone bariatric surgery and are being followed up postoperatively.

SUMMARY:
Confinement disrupts social habits, the absence of professional activity or teleworking creates the possibility for individuals to work and/or sleep at times that are most convenient for them. Investigators hypothesize that subjects with a history of obesity will tend, during confinement, to return to their spontaneous chronotype. The evolution of chronotypes between the pre-confinement period and during confinement will allow to measure the percentage of subjects who are not usually living according to their spontaneous chronotype, due to social constraints. Finally, we wish to retrospectively question the subjects on the impact of confinement on their eating habits, physical activity, mood, employment, and so on.

DETAILED DESCRIPTION:
Sleep patterns, evaluated in hunter-gatherer populations, show that without artificial interference, sleep is of course concomitant with the decrease in luminosity, but is also regulated by the outside temperature. Light pollution from night lighting and artificially regulated temperature contribute to distancing us from these physiological signals. In addition, the leisure activities linked to the screens encourage a voluntary restriction of sleep manifested by a later bedtime, whereas social constraints always impose the time of getting up. Sleep debt accumulates during the week and compensates for non-working days inducing a social jet lag of small amplitude, but repeated each week. Subjects who spontaneously or habitually develop a late chronotype (i.e. a propensity to be a "late sleeper, late riser") are the most exposed to this social jetlag between days worked when the sleep debt accumulates and days off when the sleep debt compensates.

It has been widely demonstrated that a short sleep duration promotes weight gain. Subjects with a late chronotype associate a short sleep duration on days when they work and a significant social jetlag on days when they do not work. This late chronotype is associated with unfavourable eating behaviour and more emotional eating and constitutes a risk of developing metabolic diseases.

Confinement disrupts social habits: lack of work activity or teleworking creates the possibility for individuals to work and/or sleep at times that are most convenient for them. Investigators hypothesize that subjects with a history of obesity will have tended, during confinement, to return to their spontaneous chronotype. The evolution of chronotypes between the pre-confinement period and during confinement will allow to measure the percentage of subjects who are not usually living according to their spontaneous chronotype, due to social constraints. Finally, we wish to retrospectively question the subjects on the impact of confinement on their eating habits, physical activity, mood and employment.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years-old, no upper limit)
* Included in the care pathways that prepare and then follow bariatric surgery
* Who have an e-mail address and internet access

Exclusion Criteria:

* Subjects refusing to participate
* Subjects who stayed in a country that did not organize containment during the COVID-19 pandemic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting with a medical history of obesity
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-11-02 (Estimated); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in sleep and meal schedules | before (mid-March 2020) at the end (May 11, 2020) and after containment (September 2020)

SECONDARY OUTCOMES:
Change in self-reported body weight | before (mid-March 2020) at the end (May 11, 2020) and after containment (September 2020)
Change in obesity-related quality of life evaluated by EQVOD questionnaire | before (mid-March 2020), at the end (May 11, 2020) and after confinement (September 2020).
Change in physical activity assessed by the short form of International Physical Activity Questionnaire (sf-IPAQ) | before (mid-March 2020), at the end (May 11, 2020) and after confinement (September 2020).
Change in mood and anxiety assessed by the Hospital Anxiety and Depression Scale (HADS) | before (mid-March 2020) at the end (May 11, 2020)
Change in working status | before (mid-March 2020) at the end (May 11, 2020)
Change in food security status assessed by the Household Food Security Scale Measure (HFSSM) | before (mid-March 2020), at the end (May 11, 2020) and after containment (September 2020).
Search for a correlation between evolution of the chronotype and evolution of the weight, IPAQS score, HADS score, etc. | before (mid-March 2020), at the end (May 11, 2020) and after containment (September 2020).

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Laure Borel, MD, PhD, Principal Investigator — University Hospital, Grenoble

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Borel AL. Sleep Apnea and Sleep Habits: Relationships with Metabolic Syndrome. Nutrients. 2019 Nov 2;11(11):2628. doi: 10.3390/nu11112628. PMID 31684029